CLINICAL TRIAL: NCT05500573
Title: Sex Selection of Human Spermatozoa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1306014043
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Infertility; IVF
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Sperm ejaculates are processed by an in-house protocol that utilized a multilayer density gradient comprised of four concentrations: 20%, 40%, 60%, and 90% to attempt selection of gender specific spermatozoa.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sperm sorting (Experimental): Selection of gender specific spermatozoa using a multilayer density gradient
  Interventions: Procedure: Sperm Sorting

INTERVENTIONS:
Procedure: Sperm Sorting — Selection of gender specific spermatozoa using a multilayer density gradient solution
  Other Names: Sperm Sex Selection

SUMMARY:
This study aims to demonstrate a reliable method of selecting gender specific sperm. X-bearing spermatozoa and Y-bearing spermatozoa will be identified from the density gradient layers. The selected gender specimen will then be utilized for assisted reproductive fertilization- in vitro fertilization or intrauterine insemination which are routine standard of care procedures.

DETAILED DESCRIPTION:
The study aim is to test a simple, reliable, and inexpensive method to attempt selection of gender specific spermatozoa. Couples will undergo evaluation and treatment according to the standard clinic procedures. Sperm samples provided for infertility treatment will be further analyzed routine semen analysis for volume, concentration, mobility and morphology. Sperm samples will be provided by consenting males undergoing infertility treatment. A multilayer density gradient will be performed utilizing an FDA approved solution, Enhance-S Plus Cell Isolation Media (Vitrolife, San Diego, CA).

This density gradient is also used for standard semen preparation for intrauterine insemination. X-bearing spermatozoa and Y-bearing spermatozoa will be identified from the density gradient fractions. Sperm suspensions will be smeared on slides for FISH analysis using centromeric probes for chromosomes 18, X, and Y. The ratio of X- to Y- chromosome bearing spermatozoa will be assessed as a percentage on at least 200 cells per slide. Aneuploid cells and those without signals will be omitted. Unselected fractions of each sample will serve as controls. The rate of X-bearing spermatozoa after 4-layer density gradient will be calculated. After thorough counseling, the selected preconception gender specimen will then be utilized for assisted reproductive fertilization- in vitro fertilization with or without intracytoplasmic sperm injection (ICSI) or intra uterine insemination which are routine standard of care procedures.

ELIGIBILITY:
Inclusion Criteria:

* Couples undergoing infertility treatment with IVF or insemination seeking gender specific offspring for medical and non medical reasons

Exclusion Criteria:

* Severe male factor

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2013-11-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of gender bearing spermatozoa after 4-layer density gradient | 8 years
Rate of embryos of the desired gender in couples | 8 years
Rate of offspring of the desired gender in couples | 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Gianpiero Palermo, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Center for Reproductive Medicine- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheung S, Elias R, Xie P, Rosenwaks Z, Palermo GD. A non-randomized clinical trial to determine the safety and efficacy of a novel sperm sex selection technique. PLoS One. 2023 Mar 22;18(3):e0282216. doi: 10.1371/journal.pone.0282216. eCollection 2023. PMID 36947521